CLINICAL TRIAL: NCT03200327
Title: Comparison of Anterior Vaginal Sacrospinofixation With Laparoscopic Promontofixation for the Treatment of Anterior and Apical Genitourinary Prolapse
Acronym: SAPPRO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: withdrawal of vaginal prosthesis from the market
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOIGCSMERRI/2016/RdT01; 2017-A01201-52 (Other: ANSM)
Record Dates: First submitted 2017-06-23; First posted 2017-06-27 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2022-01

CONDITIONS: Prolapse Genital

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopic promontofixation (Active Comparator)
  Interventions: Procedure: promontofixation
- Anterior vaginal sacrospinofixation (Experimental)
  Interventions: Procedure: sacrospinofixation

INTERVENTIONS:
Procedure: promontofixation — reconstruction of cystoceles using a subvesical prosthesis
  Arms: laparoscopic promontofixation
Procedure: sacrospinofixation — Utero-vaginal suspension by bilateral anterior sacrospinofixation using the vaginal route
  Arms: Anterior vaginal sacrospinofixation

SUMMARY:
The investigators anticipate a reduced risk of post-operational de novo stress urinary incontinence following surgery for vaginal sacrospinofixation, associated with reduced costs, comparable functional and anatomical efficacy and no increase in morbidity and rate of dyspareunia with the new treatment

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* Patient must be available for 12 month follow-up
* Patient is ≥50 and <80 years old
* Patient has pelvic prolapse stage 2 or above according to international POP-Q score, concerning the anterior and apical compartments, justifying surgical treatment
* Patients not having preoperational stress urinary incontinence or having mild stress urinary incontinence not causing significant functional problems (response <2 to question 17 of PFDI-20 questionnaire). It is possible that patients with hidden stress urinary incontinence will be recruited

Exclusion Criteria:

* The subject is participating in an interventional study, or is in a period of exclusion determined by a previous study
* The patient is under safeguard of justice or state guardianship
* The subject refuses to sign the consent
* Patient with communication issues preventing comprehension of information and administration of questionnaires
* Pelvic prolapse not affect anterior and apical compartments, regardless of stage
* Patient with preoperative dyspareunia (patients with mild sexual discomfort related to prolapse may be included
* Patient presents with preoperative stress urinary incontinence responsible of significant functional incapacity (response ≥2 to question 17 of PFDI-20 questionnaire).
* Indication for concomitant suburethral sling
* Patient with previous history of surgery for stress urinary incontinence
* Indication of concomitant perineorrhaphy surgery with or without myorrhaphy (in both groups).
* Contra-indication for general anesthetic
* Current urinary infection
* Current vaginal infection

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 55 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Compare the rate of de novo problematic stress urinary incontinence, operable or not, between groups response | 12 months after intervention
  ≥ 2 to question 17 of PFDI-20 questionnaire

SECONDARY OUTCOMES:
De novo dyspareunia rate the dyspareunia between groups | 12 months after the initial intervention
  ≥ 2 to question 11 of the PISQ-IR questionnaire.
Quality of sexual life between groups | 12 months after the initial intervention
  PISQ-IR questionnaire.
Re-intervention for suburethral band (BSU) in de novo SUI between groups | up to 12 months after the initial intervention
  binary: yes/no.
Compare anatomical prolapse symptoms between groups | at 6 weeks and 12 months after intervention
  POP-Q questionnaire
Compare functional prolapse symptoms between groups | at 6 weeks and 12 months after intervention
  PFDI-20 questionnaire
Compare quality of life associated to pelvic floor issues between groups | at 6 weeks and 12 months after intervention
  PFIQ questionnaire
Compare general quality of life between groups | at 6 weeks and 12 months after intervention
  SF12 questionnaire
Compare global satisfaction between groups | at 6 weeks and 12 months after intervention
  PGI-I questionnaire
Compare perioperational morbidity between groups | at 6 weeks and 12 months after intervention
  complication assessed as stage ≥2 on Clavien-Dindo classification, or according to the ICS/IUGA classification.
Compare direct and indirect costs of the 2 interventions | 12 months after intervention

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - CHU de clermont-Ferrand, Clermont-Ferrand
  - CHU de Lille, Lille
  - HFME - Hospices Civils de Lyon, Lyon
  - Clinique Beau-Soleil, Montpellier
  - CHU de Montpellier, Montpellier
  - CHU Nimes, Nîmes

REFERENCES:
- [Result] de Tayrac R, Cosson M, Panel L, Compan C, Zemmache MZ, Bouvet S, Wagner L, Fatton B, Lamblin G. Urinary and sexual impact of pelvic reconstructive surgery for genital prolapse by surgical route. A randomized controlled trial. Int Urogynecol J. 2022 Jul;33(7):2021-2030. doi: 10.1007/s00192-021-05071-8. Epub 2022 Jan 19. PMID 35044477